CLINICAL TRIAL: NCT06592183
Title: Effect of Speech Rehabilitation Based on Mobile Application for People With Dysarthria After Stroke: A Single-Center, Investigator-Blinded, Randomized, Crossover Trial
Brief Title: Speech Rehabilitation Based on Mobile Applications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Yunjung Kim, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004205
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Motor Speech Disorder
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a single-center, investigator-blinded, randomized, crossover effectiveness study. After recruitment, the participants will be randomly assigned to one of two groups: Group 1 will first receive smartphone-based speech therapy and then usual care as a control, whereas Group 2 will be on waitlist control first and then receive speech therapy. In this study, both the objective and subjective measurements will be performed three times: at baseline, post-phase 1 study (week 4), and post-phase 2 study (week 8). The study includes three intervention cycles, and for each research cycle, 12 subjects will be recruited to participate (6 per each group × 3 cycles).
Who Masked: Outcomes Assessor
Masking Description: Due to the interactive nature of rehabilitation, masking the intervention to patients and research investigators is impossible. Therefore, separate outcome assessors will be blinded, who will not be involved in the treatment procedures, to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will use a speech therapy application, a software designed for post-stroke dysarthria speech therapy and provided in the form of a mobile application. The application provides intensive speech treatment, including respiration, phonation, resonance, prosody, and articulation exercises. The system analyzes patients' voices collected while using the application and delivers the results through real-time visual and summary feedback, increasing patients' ability to self-monitor.
  Interventions: Behavioral: Smart-phone based, self-driven speech rehabilitation
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Smart-phone based, self-driven speech rehabilitation — Participants will perform the speech exercises for 60 min per day. Participants may complete the speech exercises all at once or split them into several sessions. Thus, participants assigned to the intervention group will use the application for 30-60 min daily, 5 days per week, for 4 consecutive weeks.
  Arms: Intervention

SUMMARY:
This study evaluates the efficacy of smartphone-based speech therapy administered at home compared with usual care. Participants will be randomized into the treatment and waitlist control groups with an allocation ratio of 1:1.

DETAILED DESCRIPTION:
Despite the importance of dysarthria intervention in post-stroke rehabilitation, further research in this area remains underexplored. This study builds on previous research on the use of smartphone-based dysarthria interventions based on motor learning principles, such as repetitive training and feedback and neuroplasticity through repetition, motivation, and reward. The treatment duration of 1h, 5 times a week for 4 weeks, is consistent with previous behavioral interventions for post-stroke dysarthria. This study aimed to determine whether the condition of patients with stroke can be improved through the use of smartphone-based interventions. This is a single-center, investigator-blinded, randomized, crossover effectiveness study. In this study, both the objective and subjective measurements will be performed three times: at baseline, post-phase 1 study (week 4), and post-phase 2 study (week 8). The study includes three intervention cycles, and for each research cycle, 12 subjects will be recruited to participate (6 per each group × 3 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to use a smartphone-based speech therapy application, as determined by self-reporting cognitive abilities.
* Speaks English as a native language.

Exclusion Criteria:

* Unable to use smartphone application or conduct speech assessment due to severe speech impairment.
* Self-reported co-existing progressive neurological disorders that can affect dysarthria (e.g., dementia, Pick's disease, Huntington's disease, Parkinson's disease, or Parkinsonism).
* Patient with severe mental disorders as self-reported (e.g., depression, schizophrenia, alcohol addiction, or drug addiction).
* Illiterate patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility on a visual analogue scale (VAS) | Immediately after and 8 weeks after treatment
  Speech intelligibility ratings are often estimated using a visual analogue scale . Listeners will be asked to rate the degree to which they are able to understand the speech samples using a horizontally oriented continuous scale with end points labeled, totally unintelligible and completely intelligible (0-100). The averaged score from the listeners will serve as the speech intelligibility score of the participants.

SECONDARY OUTCOMES:
Dysarthria Impact Profile (DIP) | Immediately after and 8 weeks after treatment
  DIP is an assessment tool designed to measure the psychosocial impact of dysarthria on affected individuals. It consists of several sections with statements rated on a five-point scale, ranging from "strongly agree" to "strongly disagree." DIP incorporates positively and negatively worded statements with differing scoring schemes. The fifth section prompts participants to list and rank their main concerns, including speech impairment. The final score indicates the global impact of dysarthria, with lower scores indicating a higher level of impact.
Quality of Life in the Dysarthria Speaker | Immediately after and 8 weeks after treatment
  QoL-DyS is a patient-centered measure designed to evaluate the self-perceived quality of life in individuals with post-stroke dysarthria. This measure consists of 40 items, each rated on a scale of 0 (never) to 4 (all of the time). The questionnaire is divided into 4 parts, with 10 questions each, covering the following aspects: speech characteristics, situational difficulty, compensatory strategies, and perceived reactions of others.
Carer Communication Outcomes After Stroke (CaCOAST) | Immediately after and 8 weeks after treatment
  CaCOAST assesses the carer's perception of the patient's communication effectiveness and its impact on their quality of life. The measure has 20 items, each assessed on a scale of 0 to 4, and a percentage summary measure is calculated. The first 15 items assess the carer's perception of the patient's communication, whereas the last 5 assess the impact of the patient's communication difficulties on the carer's quality of life.
Speaking Rate (syl/s) | Immediately after and 8 weeks after treatment
  Changes in acoustic signals will be measured. Specifically, changes in the number of syllables per second (speaking rate) will be reported as slow speaking rate is a frequent speech characteristic of people with stroke.
Acoustic vowel space (KHz) | Immediately after and 8 weeks after treatment
  Changes in acoustic signals will be measured. Specifically, changes in the size of acoustic vowel space (in KHz2) will be reported, as this is well known to be reduced in speakers with stroke and to correlate with speech intelligibility.

OTHER OUTCOMES:
System Usability Scale (SUS) | Immediately after and 8 weeks after treatment
  SUS is a 10-item questionnaire (usability performance in the aspects of effectiveness, efficiency, and overall ease of use) with 5 response options for respondents, from strongly agree to strongly disagree. For the interpretation of the results, the scores are normalized and converted into a total score of 100. Based on research, a SUS score above 68 would be considered above-average usability, and above 80.3 would be considered excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Jinwoo Kim, PhD, Study Director — Haii Corp.
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the data which will be collected (including voice), the investigators do not plan to share IPD with other researchers.